CLINICAL TRIAL: NCT00979576
Title: A Phase I/II Study of Continuous, Concomitant Oral Treatment With BIBF 1120 and Pemetrexed - a Phase I, Open-label, Dose-escalation Study & a Phase II, 2 Arm, Randomized, Double-blind, Placebo-controlled Study in Japanese Patients With Stage IIIB/IV or Recurrent Non-small-cell Lung Cancer After Failure of Chemotherapy
Brief Title: BIBF 1120 in Combination With Pemetrexed in Advanced Non Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.28
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

ARMS (3):
- BIBF 1120 BID + Pemetrexed (Experimental): Phase I part: Find MTD by using low, medium or high BIBF 1120 twice daily and 500mg/m^2 pemetrexed once every 3 weeks
  Interventions: Drug: BIBF 1120 M + Pemetrexed; Drug: BIBF 1120 H + Pemetrexed; Drug: BIBF 1120 L + Pemetrexed
- BIBF 1120 BID (RD) + Pemetrexed (Experimental): PHase II part: Study arm
  Interventions: Drug: BIBF 1120 RD + Pemetrexed
- BIBF 1120 BID(Placebo) + Pemetrexed (Experimental): Phase II part: Comparator arm
  Interventions: Drug: BIBF 1120 Placebo + Pemetrexed

INTERVENTIONS:
Drug: BIBF 1120 M + Pemetrexed — BIBF 1120 medium dose bid+ Pemetrexed 500 mg/m^2
  Arms: BIBF 1120 BID + Pemetrexed
Drug: BIBF 1120 H + Pemetrexed — BIBF 1120 high dose bid+ Pemetrexed 500 mg/m^2
  Arms: BIBF 1120 BID + Pemetrexed
Drug: BIBF 1120 RD + Pemetrexed — confirmed dose of BIBF 1120 bid + Pemetrexed 500 mg/m^2
  Arms: BIBF 1120 BID (RD) + Pemetrexed
Drug: BIBF 1120 L + Pemetrexed — BIBF 1120 low dose bid+ Pemetrexed 500 mg/m^2
  Arms: BIBF 1120 BID + Pemetrexed
Drug: BIBF 1120 Placebo + Pemetrexed — placebo BIBF 1120 bid + Pemetrexed 500 mg/m^2
  Arms: BIBF 1120 BID(Placebo) + Pemetrexed

SUMMARY:
The objectives of this trial are to estimate the following in Japanese patients with advanced NSCLC of stage IIIB/IV or with recurrence after failure of first-line chemotherapy.

Phase I part The objective of the phase I part is to define the Maximum Tolerated Dose (MTD) of BIBF 1120 at a dose level up to twice daily 200 mg with standard dose of pemetrexed (500 mg/m^2) and to determine the Recommended Dose (RD) for the phase II part.

Phase II, to investigate the efficacy and safety of BIBF 1120 in combination with pemetrexed (500 mg/m^2) as compared to pemetrexed (500 mg/m^2) + placebo

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients of age >=20 and <=74 years at informed consent
2. Histologically or cytologically confirmed, Non Small Cell Lung Cancer (NSCLC) of stage IIIB or IV or recurrent NSCLC
3. Relapse or failure of 1 first-line prior chemotherapy
4. Life expectancy of at least 3 months
5. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
6. Patients who have sufficient baseline organ function over 4 weeks and whose laboratory data meet the following criteria at the enrolment

   * Haemoglobin >=9.0 g/dL
   * Absolute neutrophil count (ANC) >=1500/mm^3
   * Platelet count >=100 000/mm^3
   * Total bilirubin under the upper limit of normal
   * AST/SGOT and/or ALT/GPT <=1.5 x upper limit of normal (if related to liver metastases <=2.5 x upper limit of normal also)
   * Proteinuria Common Terminology Criteria for Adverse Events (CTCAE) grade 1 or less
   * Calculated creatinine clearance by Cockcroft Gault >=45 mL/min
   * Prothrombin time-international normalized ratio (PT-INR) and/or partial thromboplastin time (PTT) greater than 50% deviation from normal limits
   * arterial oxgen pressure (PaO2) >=60 torr or oxygen saturation by pulse-oximeter SpO2 >=92%
7. Patient has given written informed consent which must be consistent with ICH-GCP and local legislation.

Exclusion criteria:

1. Patients who have received treatment with other investigational drugs or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with this trial or who have not recovered from side effects of such therapy (except for alopecia)
2. Patients who have received chemo-, hormone-, immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 4 weeks prior to treatment with the trial drug or who have not recovered from side effects of such therapy (except for alopecia) .
3. Patients who have received radiotherapy within the following period Phase I part: the past 4 weeks prior to treatment with the trial drug (in case of palliative radiotherapy such as for extremities, within the past 2 weeks prior to treatment with the trial drug)
4. Previous therapy with other vascular endothelial growth factor receptor (VEGFR) inhibitors or vascular endothelial growth factor (VEGF) ligand inhibitors for treatment of NSCLC
5. Previous therapy with BIBF 1120 and/or pemetrexed for treatment of NSCLC and any contraindications for therapy with pemetrexed
6. Patients who have active brain metastases
7. Leptomeningeal disease
8. Patients with distinct or suspected pulmonary fibrosis or interstitial lung disease by the CT findings, or patients with a previous history of pulmonary fibrosis or interstitial lung disease (except irradiation-pneumonitis appearing radiation field with past radiotherapy).
9. Radiographic evidence of cavitary or necrotic tumors
10. Centrally located tumors with radiographic evidence (CT or MRI) of local invasion of major blood vessels
11. History of clinically significant haemoptysis within the past 3 months
12. History of major thrombotic or clinically relevant major bleeding event in the past 6 months
13. Known inherited predisposition to bleeding or thrombosis
14. Significant cardiovascular diseases
15. Significant weight loss (>10%) within the past 6 weeks prior to treatment in the present trial
16. Current peripheral neuropathy CTCAE grade 2 or greater except due to trauma
17. Pre-existing ascites and/or clinically significant pleural effusion
18. Major injuries and/or surgery within the past 4 weeks prior to randomisation with incomplete wound healing
19. Clinically serious infections
20. Decompensated diabetes mellitus
21. Contraindication to high dose steroid therapy
22. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
23. Patients who have active or chronic hepatitis C and/or B infection and diagnosis of human immunodeficiency virus (HIV) infection
24. Other malignancy other than basal cell skin cancer, carcinoma in situ or intra-mucosal cancer that were judged to be cured by adequate treatment and disease-free interval is more than 5 years
25. History of serious drug hypersensitivity
26. Serious illness or concomitant non-oncological disease such as neurologic-, psychiatric-, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation
27. Therapeutic anticoagulation (except low dose heparin and/or heparin flush as needed for maintenance of an indwelling intravenous device) or antiplatelet therapy
28. Patients who are sexually active and unwilling to use a medically acceptable method of contraception
29. Pregnancy or breast feeding
30. Active alcohol or drug abuse
31. Patients unable to comply with the protocol
32. Other patients judged ineligible for enrolment in the study by the investigator or subinvestigator.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-10-16 (Actual); Primary Completion 2015-02-16 (Actual); Study Completion 2015-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Japan (3):
  - 1199.28.003 Boehringer Ingelheim Investigational Site, Chiba,Kashiwa
  - 1199.28.002 Boehringer Ingelheim Investigational Site, Miyakojima-ku, Osaka
  - 1199.28.001 Boehringer Ingelheim Investigational Site, Osaka-Sayama, Osaka

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Daga H, Takeda K, Okada H, Miyazaki M, Ueda S, Kaneda H, Okamoto I, Yoh K, Goto K, Konishi K, Sarashina A, Tanaka T, Kaiser R, Nakagawa K. Phase I study of nintedanib in combination with pemetrexed as second-line treatment of Japanese patients with advanced non-small cell lung cancer. Cancer Chemother Pharmacol. 2015 Dec;76(6):1225-33. doi: 10.1007/s00280-015-2896-3. Epub 2015 Nov 11. PMID 26560486
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 patients were enrolled in the study however one patient did not meet the inclusion criteria and therefore did not participate in the study.
Groups:
- BIBF 1120 100 mg + Pemetrexed 500 mg/m^2: Treatments were administered in 21 day courses. Patients received pemetrexed 500 mg/m^2 administered by intravenous infusion on day 1 and BIBF 1120 (nintedanib) 100 mg administered orally once on day 2 and twice daily (b.i.d.) from day 3 to day 21 in cycle 1 and b.i.d. from day 2 to day 21 in further cycles. In case that a patient had to discontinue pemetrexed, the patient was allowed to continue nintedanib monotherapy if the patient had been treated with the nintedanib combination therapy with pemetrexed for at least 4 courses.
- BIBF 1120 150 mg + Pemetrexed 500 mg/m^2: Treatments were administered in 21 day courses. Patients received pemetrexed 500 mg/m^2 administered by intravenous infusion on day 1 and BIBF 1120 (nintedanib) 150 mg administered orally once on day 2 and twice daily (b.i.d.) from day 3 to day 21 in cycle 1 and b.i.d. from day 2 to day 21 in further cycles.
  In case that a patient had to discontinue pemetrexed, the patient was allowed to continue nintedanib monotherapy if the patient had been treated with the nintedanib combination therapy with pemetrexed for at least 4 courses.
- BIBF 1120 200 mg + Pemetrexed 500 mg/m^2: Treatments were administered in 21 day courses. Patients received pemetrexed 500 mg/m^2 administered by intravenous infusion on day 1 and BIBF 1120 (nintedanib) 200 mg administered orally once on day 2 and twice daily (b.i.d.) from day 3 to day 21 in cycle 1 and b.i.d. from day 2 to day 21 in further cycles.
  In case that a patient had to discontinue pemetrexed, the patient was allowed to continue nintedanib monotherapy if the patient had been treated with the nintedanib combination therapy with pemetrexed for at least 4 courses.
Period: Combination Treatment Phase
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2
Started | 3 | 6 | 9
Completed | 0 | 0 | 0
Not Completed | 3 | 6 | 9
Not completed — Progressive disease | 3 | 1 | 5
Not completed — Dose limiting toxicity | 0 | 3 | 2
Not completed — Adverse Event | 0 | 2 | 2
Period: Combination Followed by Monotherapy
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2
Started | 0 | 2 | 1
Completed | 0 | 0 | 0
Not Completed | 0 | 2 | 1
Not completed — Progressive Disease | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Treated set: all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2 | Total
Number analyzed (Participants) | 3 | 6 | 9 | 18
Age, Continuous [Median (Full Range); unit: years] | 61.0 [60 to 66] | 66.0 [54 to 70] | 64.0 [30 to 70] | 64.0 [30 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 2 | 4 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities
Description: Number of participants with dose limiting toxicity (DLT) in combination therapy of BIBF 1120 and pemetrexed during the first course
Time Frame: During the first course, 21 days
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 3 | 6 | 9
Participants | 0 | 1 | 2

2. Primary Outcome: Adverse Events According to Common Terminology Criteria for Adverse Events (CTCAE), Version 3.0 for All Courses
Description: Number of patients with adverse events according to worst Common Terminology Criteria for Adverse Events (CTCAE), version 3.0 for all courses.
  CTCAE grades are: 1 (mild AE), 2 (moderate AE), 3 (severe AE), 4 (life-threatening or disabling AE) or 5 (death related to AE).
Time Frame: Between first administration of pemetrexed and 28 days after last administration of pemetrexed and/or BIBF 1120, up to 1020 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 3 | 6 | 9
participants
  Grade 1 | 0 | 0 | 1
  Grade 2 | 2 | 1 | 2
  Grade 3 | 1 | 5 | 5
  Grade 4 | 0 | 0 | 1
  Grade 5 | 0 | 0 | 0

3. Secondary Outcome: Overall Response Rate
Description: Number of participants with complete response (CR) or partial response (PR) according to the Response Evaluation Criteria In Solid Tumors (RECIST) 1.0
Time Frame: Every 6 weeks after start of study treatment until end of treatment, up to 992 days
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 3 | 6 | 9
Participants
  Complete response | 0 | 0 | 0
  Partial response | 0 | 1 | 1

4. Secondary Outcome: Disease Control Rate
Description: Number of participants with complete response (CR), partial response (PR) or stable disease (SD) according to the Response Evaluation Criteria In Solid Tumors (RECIST) 1.0
Time Frame: Every 6 weeks after start of study treatment until end of treatment, up to 992 days
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 3 | 6 | 9
Participants | 2 | 4 | 6

5. Secondary Outcome: Duration of Disease Control
Description: Duration of disease control was defined as the time period from the first study drug administration to the progressive disease (PD) or death of patients, whichever occurred earlier.
Time Frame: From first study drug administration until PD or death, up to 1003 days
Population: Patients from the treated set who achieved disease control
Measure: Median (Full Range); unit: Days
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 2 | 4 | 6
Days | 248.5 [162 to 335] | 228.5 [168 to 587] | 149.0 [121 to 1003]

6. Secondary Outcome: Number of Participants With Clinically Relevant Abnormalities in Laboratory Parameters
Description: Number of participants with clinically relevant abnormalities in laboratory parameters reported as adverse events which occurred in >= 20% of patients
Time Frame: as for outcome 2
Population: Treated set
Measure: Number; unit: participants
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 3 | 6 | 9
participants
  Alanine aminotransferase increased | 2 | 6 | 8
  Gamma-glutamyltransferase increased | 2 | 5 | 8
  Aspartate aminotransferase increased | 2 | 5 | 7
  Lymphocyte count decreased | 2 | 1 | 2
  Neutrophil count decreased | 2 | 3 | 4
  White blood cell count decreased | 2 | 2 | 3
  Blood alkaline phosphatase increased | 0 | 1 | 4
  Blood albumin decreased | 0 | 1 | 3
  Haemoglobin decreased | 1 | 1 | 3

7. Secondary Outcome: AUC0-inf of Nintedanib
Description: Area under the concentration-time curve of nintedanib in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf)
Time Frame: 5 minutes (min) before nintedanib administration and 1h, 2h, 3h, 4h, 6h, 7h, 10h and 23h 55min after nintedanib administration in cycle 1
Population: Pharmacokinetic (PK) set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 3 | 6 | 9
ng*h/mL | 105 (25.5) | 232 (60.5) | 323 (28.8)

8. Secondary Outcome: Cmax of Nintedanib
Description: Maximum measured concentration of nintedanib in plasma (Cmax)
Time Frame: as for outcome 7
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2
Number analyzed (Participants) | 3 | 6 | 9
ng/mL | 20.5 (31.0) | 37.9 (71.7) | 55.1 (29.6)

9. Secondary Outcome: AUC0-inf of Pemetrexed
Description: Area under the concentration-time curve of pemetrexed in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf)
Time Frame: 5 minutes (min) before pemetrexed administration and 10min, 40min, 1 hour (h), 2h, 4h, 6h, 23h 55min, 47h 55min after pemetrexed administration in cycles 1 and 2
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Pemetrexed 500 mg/m2: Pemetrexed 500 mg/m2 administered by intravenous infusion taken in combination with oral administration of BIBF 1120 100mg, 150mg or 200mg b.i.d..
Arm/Group | Pemetrexed 500 mg/m2
Number analyzed (Participants) | 18
ng*h/mL
  Cycle 1 | 194000 (19.9)
  Cycle 2 (N=11) | 200000 (15.9)

10. Secondary Outcome: Cmax of Pemetrexed
Description: Maximum measured concentration of pemetrexed in plasma (Cmax)
Time Frame: as for outcome 9
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Pemetrexed 500 mg/m2
Number analyzed (Participants) | 18
ng/mL
  Cycle 1 | 139000 (16.5)
  Cycle 2 (N=11) | 149000 (15.4)

ADVERSE EVENTS:
Time Frame: Between first administration of pemetrexed and 28 days after last administration of pemetrexed and/or BIBF 1120, up to 1020 days
Arm/Group | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/6 | 1/9
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 (N=3) | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 (N=6) | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2 (N=9)
Fatigue (General disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIBF 1120 100 mg + Pemetrexed 500 mg/m^2 (N=3) | BIBF 1120 150 mg + Pemetrexed 500 mg/m^2 (N=6) | BIBF 1120 200 mg + Pemetrexed 500 mg/m^2 (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 7
Glossitis (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 4
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4
Face oedema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 4 | 1
Influenza like illness (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 4
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 6 | 8
Aspartate aminotransferase increased (Investigations) | 2 | 5 | 7
Blood albumin decreased (Investigations) | 1 | 1 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood calcium increased (Investigations) | 1 | 0 | 0
Blood chloride increased (Investigations) | 0 | 1 | 0
Blood creatine increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 1 | 1 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 5 | 8
Glucose urine present (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 3
Lymphocyte count decreased (Investigations) | 2 | 1 | 2
Neutrophil count decreased (Investigations) | 2 | 3 | 4
Neutrophil count increased (Investigations) | 0 | 2 | 0
Platelet count decreased (Investigations) | 0 | 1 | 1
Thyroxine free increased (Investigations) | 1 | 0 | 0
Tri-iodothyronine free decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 2 | 2 | 3
White blood cell count increased (Investigations) | 1 | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Convulsion (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 4
Proteinuria (Renal and urinary disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 3
Flushing (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The trial was planned to comprise of two parts, with the phase II being based on the results of another study. The other study was stopped early due to futility analysis therefore only phase I of the study was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.